CLINICAL TRIAL: NCT02539654
Title: An Open-Label, Single-Dose, Pharmacokinetic Study of EXE844 Sterile Otic Suspension, 0.3% in Pediatric Subjects Following Tympanostomy Tube Surgery
Brief Title: Pediatric Pharmacokinetic (PK) Study of EXE844 Otic Suspension in Otitis Media at the Time of Tympanostomy Tube Insertion (OMTT)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EXE844b-C003
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2017-11

CONDITIONS: Otitis Media With Effusion in Children; Otitis Media Recurrent
MeSH Terms: interventions — Middle Ear Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EXE844 (Experimental): EXE844 Sterile Otic Suspension, 0.3%, single ototopical dose (4 drops) in each ear following tympanostomy tube insertion
  Interventions: Drug: EXE844 Sterile Otic Suspension, 0.3%; Procedure: Tympanostomy Tube Insertion

INTERVENTIONS:
Drug: EXE844 Sterile Otic Suspension, 0.3%
Procedure: Tympanostomy Tube Insertion

SUMMARY:
The purpose of this study is to describe the pharmacokinetics (PK) of EXE844 Sterile Otic Suspension, 0.3% following a single bilateral ototopical dose in pediatric subjects, immediately after bilateral tympanostomy tube surgery.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent acute otitis media (RAOM) or chronic otitis media with effusion (COME) and eligible for bilateral myringotomy and tympanostomy tube insertion;
* Legally Authorized Representative (LAR) must read and sign the informed consent;
* Parent or caregiver must agree to complete the required study visits and comply with the requirements of the study;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Menarcheal females;
* Previous otologic or otologic-related surgery within the past 30 days or ongoing complications;
* Existing perforation of the eardrum;
* Current acute otitis externa (AOE), malignant otitis externa (MOE) or other conditions which could interfere with evaluation of the study drug;
* Any systemic disease or disorder, complicating factor or structural abnormality that would negatively affect the conduct or outcome of the study;
* Use of prohibited medications or inadequate washout of any medication including systemic and topical antibiotics, steroids and/or analgesics;
* Weighs less than 8 kg;
* Other protocol-specified exclusion criteria may apply.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2016-06-24 (Actual); Study Completion 2016-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, GCRA, Pharma, Study Director — Alcon Research
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2 investigational sites located in the US.
Pre-assignment Details: All 14 enrolled participants were treated. This reporting group includes all enrolled participants (14).
Period: Overall Study
Arm/Group | EXE844
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all participants who had tympanostomy tubes (TT) inserted, received a dose of study drug, had at least 1 plasma sample following study drug exposure, and had no collection or analytical deviations affecting the integrity of the pharmacokinetic (PK) data (PK Analysis Set).
Arm/Group | EXE844
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.4 (2.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Maximum Analyte Plasma Concentration (Cmax)
Description: Based on serum samples collected at pre-determined nominal time points, dependent on observed concentrations. EXE844 (AL-60371) concentration values below the lower limit of quantification (<0.05 ng/mL) were replaced by one-half the lower limit of quantification in the calculation of the summary statistics. Similarly for EXE844 glucuronide metabolite (AL-91591), concentration values below the lower limit of quantification (<0.5 ng/mL) were replaced by one-half the lower limit of quantification in the calculation of the summary statistics.
Time Frame: Day 1, pre-dose 0 hour (up to 30 minutes prior to dose), 0.5, 1, 2, 4, 6 hours post-dose
Population: PK analysis set, with at least 1 post-dose quantifiable plasma concentration for each individual analyte [EXE844 (AL-60371) and EXE844 glucuronide metabolite (AL-91591)]
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | EXE844
Number analyzed (Participants) | 14
ng/mL
  AL-60371 | 2.44 (2.411)
  AL-91591: number analyzed (Participants) | 7
  AL-91591 | 1.61 (1.141)

2. Primary Outcome: Time to Reach Maximum Concentration (Tmax)
Description: as for outcome 1
Time Frame: Day 1, pre-dose 0 hour (up to 30 minutes prior to dose), 0.5, 1, 2, 4, 6 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | EXE844
Number analyzed (Participants) | 14
hours
  AL-60371 | 0.59 [0.48 to 2.1]
  AL-91591: number analyzed (Participants) | 7
  AL-91591 | 1.00 [0.55 to 2.17]

3. Primary Outcome: Area Under the Plasma Concentration-time Curve to the Last Quantifiable Sampling Time Point (AUC0-last)
Description: as for outcome 1
Time Frame: Day 1, pre-dose 0 hour (up to 30 minutes prior to dose), 0.5, 1, 2, 4, 6 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | EXE844
Number analyzed (Participants) | 9
ng*h/mL
  AL-60371 | 8.66 (6.406)
  AL-91591: number analyzed (Participants) | 7
  AL-91591 | 3.94 (4.136)

4. Primary Outcome: Area Under the Concentration-time Curve From 0 to Infinity (AUC0-inf)
Description: as for outcome 1
Time Frame: Day 1, pre-dose 0 hour (up to 30 minutes prior to dose), 0.5, 1, 2, 4, 6 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | EXE844
Number analyzed (Participants) | 8
ng*h/mL
  AL-60371 | 10.60 (7.764)
  AL-91591: number analyzed (Participants) | 1
  AL-91591 | 19.90 (NA) — Unable to compute estimate

5. Primary Outcome: Time to Last Measurable Concentration (Tlast)
Description: as for outcome 1
Time Frame: Day 1, pre-dose 0 hour (up to 30 minutes prior to dose), 0.5, 1, 2, 4, 6 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | EXE844
Number analyzed (Participants) | 11
hours
  AL-60371 | 5.90 [1.08 to 6.1]
  AL-91591: number analyzed (Participants) | 7
  AL-91591 | 2.17 [1 to 5.95]

6. Primary Outcome: Terminal Elimination Half-life (T1/2)
Description: as for outcome 1
Time Frame: Day 1, pre-dose 0 hour (up to 30 minutes prior to dose), 0.5, 1, 2, 4, 6 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | EXE844
Number analyzed (Participants) | 8
hours
  AL-60371 | 2.05 (0.821)
  AL-91591: number analyzed (Participants) | 1
  AL-91591 | 4.42 (NA) — Unable to compute estimate

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of a subject's participation in the study (up to 20 days). AE reporting began after parent/legally authorized representative (LAR) signed informed consent and if applicable, after participant signed assent. AEs are reported as pre-treatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. AEs were obtained as solicited comments from the study participants and as observations by the Investigator as outlined in the study protocol.
Groups:
- Pre-treatment: All subjects who consented to participate in the study prior to the initiation of study treatment
- EXE844: All participants who had TT inserted and received a dose of test article
Arm/Group | Pre-treatment | EXE844
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.